CLINICAL TRIAL: NCT06450899
Title: Prochlorperazine Maleate Versus Placebo for the Prophylaxis of Acute Mountain Sickness
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Colorado, Denver (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 23-0958
Record Dates: First submitted 2024-05-28; First posted 2024-06-10 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Acute Mountain Sickness
MeSH Terms: conditions — Altitude Sickness | interventions — Prochlorperazine

STUDY DESIGN:
Intervention Model Description: Prospective double-blind, placebo controlled randomized controlled trial
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: This study will be a placebo-controlled, double blinded trial. Intervention and placebo are non-identical though very similar in appearance and will be stored in opaque vials. A non-blinded study team member will be solely in charge of dispensing medications.
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Prochlorperazine Maleate (Experimental): This arm will be the interventional/experimental arm receiving prochlorperazine maleate, further described in experimental arm section.
  Interventions: Drug: Prochlorperazine Maleate
- Placebo (Placebo Comparator): The placebo arm individuals will receive a non-identical placebo.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Prochlorperazine Maleate — Currently, prochlorperazine maleate is approved by the FDA for the treatment of nausea and vomiting, and additionally used off-label as an acute migraine treatment. The FDA has approved the dose of 5-10 mg to be taken orally 3-4 times a day. The study intervention will be obtained from Belmar Pharma solutions. Individuals randomized into the study arm will receive generic prochlorperazine maleate 10 mg orally taken three times daily for one day. Participants will convene in the morning of the trial date at low altitude, where they will receive their first dose. They will then be driven to Summit Lake and break for lunch, where they will receive their second dose approximately 6 hours later. They will then hike to the summit and receive their final dose in the evening, approximately another 6 hours later.
  Other Names: Compazine
  Arms: Prochlorperazine Maleate
Drug: Placebo — The placebo arm individuals will receive a non-identical inert generic placebo tablet containing microcrystalline cellulose provided by Belmar Pharma Solutions. Placebo tablets will be taken at the same time and frequency as the study intervention drug.
  Arms: Placebo

SUMMARY:
This study is a trial looking at a drug to help prevent acute mountain sickness. The drug is prochlorperazine, a drug commonly used to treat nausea vomiting and headache. Participants will either take the drug or a placebo, and hike to and sleep at the summit of Mount Blue Sky located at 4,348 meters (14,265 feet).

DETAILED DESCRIPTION:
This study will be a double-blind randomized controlled trial to investigate the utility of prochlorperazine maleate versus placebo for the chemoprophylaxis of acute mountain sickness on rapid ascent to 4,348 meters, specifically the summit of Mount Blue Sky in the Mount Blue Sky Wilderness. Participants will be evaluated for AMS utilizing the 2018 LLQ both the evening of and morning after ascent. The primary outcome will be the presence of AMS, defined by a 2018 LLQ score equal to or greater than 3, including the presence of a headache at any measured point during the study. Individuals will convene the morning of the study in Golden, Colorado where they will receive breakfast and either placebo or prochlorperazine. They will then be driven to Summit Lake where they will break for lunch and receive the second dose of placebo or prochlorperazine. They will then hike to the Mount Blue Sky summit where they will receive their third and final dose of either placebo or intervention, spend the night in the structures at the summit, and be assessed for AMS via LLQ. In the morning, they will be assessed for AMS again, receive breakfast, and then be driven back to the original meeting point. They will be monitored by Emergency Physicians at all points during the study.

ELIGIBILITY:
Inclusion Criteria:

* Adults >18 years old.

Exclusion Criteria:

* Individuals <18 years old or >75 years old
* Pregnant women
* Individuals who reside at or have slept at elevations >1,800 meters in the last two weeks
* Individuals having taken acetazolamide, steroids, ibuprofen, anti-emetics or additional analgesics within the last 24 hours prior to study initiation
* Individuals requiring supplemental baseline oxygen or with chronic disorders known to be significantly impacted by hypoxia
* Individuals with known allergies to prochlorperazine or phenothiazines
* Individuals taking medications with significant medication interactions with prochlorperazine: Dofetilide, potassium acid phosphate, potassium chloride, potassium citrate, potassium phosphate, Yohimbe.
* Individuals with a history of dementia
* Individuals who lack decision making capacity

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 57 (Actual)
Dates: Start 2024-08-05 (Actual); Primary Completion 2024-08-28 (Actual); Study Completion 2024-08-28 (Actual)

PRIMARY OUTCOMES:
Acute Mountain Sickness | The primary outcome will be assessed during the discreet roughly 36 hour trial period. LLQs will be administered the evening of and morning after arrival to peak altitude, or at any point of self reported altitude illness.
  The primary outcome will be the presence of AMS, defined by a 2018 Lake Louise Questionnaire (LLQ) score of equal to or greater than 3, including the presence of a headache at any measured point during the study.

CONTACTS AND LOCATIONS:
Overall Officials: Elan Small, MD, Study Director — University of Colorado, Denver
Locations (1):
- Mount Blue Sky, Evergreen, Colorado, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Small E, Goldberg E, Musi M, Strickland B, Paterson R, Phillips C, Keyes LE. Prochlorperazine maleate versus placebo for the prevention of acute mountain sickness: study protocol for a randomized controlled trial. Trials. 2024 Nov 21;25(1):785. doi: 10.1186/s13063-024-08592-x. PMID 39574186

DOCUMENTS (1):
  • Informed Consent Form (2024-05-05): https://cdn.clinicaltrials.gov/large-docs/99/NCT06450899/ICF_000.pdf